CLINICAL TRIAL: NCT04167033
Title: Study of Ventricular Repolarization in Patients With Premature Ovarian Insufficiency and Influence of Estrogen-progestin Replacement Therapy
Brief Title: Ventricular Repolarization in Patients With Premature Ovarian Insufficiency (QTIOP)
Acronym: QTIOP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: APHP180160; 2019-A01002-55 (Registry Identifier: IDRCB)
Record Dates: First submitted 2019-09-26; First posted 2019-11-18 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Premature Ovarian Insufficiency
Keywords: Premature ovarian insufficiency; QTc; Torsade de pointe; Hormone replacement therapy
MeSH Terms: conditions — Primary Ovarian Insufficiency; Torsades de Pointes | interventions — Electrocardiography

STUDY DESIGN:
Intervention Model Description: This is a bicentric case-control study: 60 patients with POI followed in the endocrinology department, and 60 healthy volunteers matched with POI's patients on age (+/- 5 years), on BMI classes (BMI<18, 18-25, 25-30, 30-35, 35-40, >40) and with regular cycles (26 to 32 days).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Premature ovarian insufficiency (Experimental): 60 patients with POI followed in the endocrinology department
  Interventions: Drug: Hormone replacement therapy:effect on ventricular repolarization
- healthy volunteers (Other): 60 healthy volunteers matched with POI's patients
  Interventions: Diagnostic Test: ECG

INTERVENTIONS:
Drug: Hormone replacement therapy:effect on ventricular repolarization — Hormone replacement therapy and QTc measurement
  Arms: Premature ovarian insufficiency
Diagnostic Test: ECG — QTc measurement
  Arms: healthy volunteers

SUMMARY:
Ventricular repolarization, measured by corrected QT interval (QTc), is influenced by sex hormones. A QTc above 460msec predisposes to the risk of "torsades-de-pointes"(TdP). The investigators have recently shown that estradiol determines an increase in QTc elongation and progesterone shortens it. In addition, high gonadotropin levels (FSH or LH) are associated with QTc prolongation. Hypergonadotropic hypogonadisms (low progesterone and high gonadotropins) are therefore hormonal situations that promote QTc prolongation. Premature ovarian insufficiency (POI) is one of them. Its management is based on the prescription of hormone replacement therapy (HRT). Epidemiological studies have shown that these patients would be at increased risk of cardiovascular mortality. Our team is interested in the effect of this pathological hormonal situation and its HRT on ventricular repolarization in order to define whether this is a population at risk for long QTc.

DETAILED DESCRIPTION:
Ventricular repolarization, measured by the duration of the heart rate corrected QT interval (QTc), is influenced by sex hormones. A QTc above 460msec predisposes to the risk of torsades-de-pointes (TdP); ventricular arrhythmias that can lead to sudden death.

From puberty to menopause, QTc is longer in women than in men (~10-15msec difference) and varies in women according to the menstrual cycle (~5-10msec). This explains the increased risk of TdP in women compared to men. During the menstrual cycle, the risk is highest for women during the follicular phase compared to the luteal phase. The investigators have recently shown that estradiol determines an increase in QTc elongation and progesterone shortens it. In addition, high gonadotropin levels (FSH or LH) are associated with QTc prolongation. Hypergonadotropic hypogonadisms (low progesterone and high gonadotropins) are therefore hormonal situations that promote QTc prolongation.

Premature ovarian insufficiency (POI) affects 1% of women under 40 years of age and is characterized by hypergonadotropic hypogonadism. POI is associated with hormonal deficiencies responsible for amenorrhea and infertility. Management is based on the prescription of hormone replacement therapy (HRT). Epidemiological studies have shown that these patients would be at increased risk of cardiovascular mortality. HRT will be based on the combination of an estrogen and a progestin and will lead to a variable decrease in gonadotropins, depending on the steroid hormones/doses used. Our team, after structuring one of the largest international cohorts of patients with POI, is interested in the effect of this pathological hormonal situation and its HRT on ventricular repolarization to define whether this is a population at risk for long QTc. Indeed, ECG follow-up is recommended and many drugs (cardiovascular or not), are to be avoided, or even contraindicated in situations at risk of long QTc.

ELIGIBILITY:
Inclusion Criteria:

Patients with POI

* Patient aged 18 to 41 years
* Patient with POI diagnostic criteria (FSH >25UI/l twice at intervals of a few weeks) with amenorrhea
* No hormone treatment interacting with the gonadotropic axis for at least one month before inclusion
* Patient who has signed informed consent
* Patient affiliated to a social security system

Healthy volunteers (including POI control group)

* Healthy women, aged 18 to 40 years, age-matched (+/- 5 years), and by BMI class (BMI<18, 18-25, 25-30, 30-35, 35-40, >40) compared to women with BPI
* Women with regular cycles of 26 to 32 days
* Women who has signed an informed consent form
* Patient affiliated to a social security system

Exclusion Criteria:

Patients with POI

* Patient on HRT during the 1st evaluation
* Pregnant or breastfeeding woman
* Treatment regimen known to lengthen QT or act on ventricular repolarization
* Cardiac history in particular cardiac rhythm disorder
* Diabetes
* Patient on AME (unless derogation from affiliation),
* Severe renal insufficiency (MDRD <30ml/min/m²)

Healthy volunteers (including POI control group)

* Diabetes or any chronic disease (including cardiovascular and endocrine)
* Pregnant or breastfeeding woman
* Hormonal contraceptive treatment in progress or stopped less than 3 months ago
* Chronic treatment affecting the duration of QTc
* Woman under AME (unless affiliation derogation)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2021-04-14 (Actual); Primary Completion 2027-04-13 (Estimated); Study Completion 2027-06-13 (Estimated)

PRIMARY OUTCOMES:
Duration of QTc | in the luteal phase between Day22 and Day25
  Compare the duration of QTc in patients with non-substituted POI with that of matched healthy volunteers on cardiovascular risk factors. The QTc will be measured by the Fridericia method

SECONDARY OUTCOMES:
Duration of QTc | the day before and between Day22 and Day60 after the introduction of HRT
  Measure the duration of QTc in women with POI before and after the introduction of HRT
Duration of QTc | in the luteal phase between Day22 and Day25
  Study the association between sex hormone levels (gonadotropins, steroid hormones) and QTc duration, as well as their variation in patients with POI and healthy volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Anne Bachelot, Pr, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Joe Elie Salem, MD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (3):
- France (3):
  - Hopital Haut Leveque, Bordeaux
  - BACHELOT, Paris
  - Pitié Salpêtrière, Paris